CLINICAL TRIAL: NCT06721845
Title: Non-Cirrhotic Hyperammonemia Versus Hyperlactatemia in Septic Patients and Impact of Treatment
Status: Completed | Type: Observational
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, ashraf magdy eskandr, professor of anesthesia, ICU, Pain Management, Menoufia University
Other Study IDs: 6/2023, ANET40
Record Dates: First submitted 2024-11-29; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Sepsis
Keywords: sepsis; hyperammonemia; hyperlactemia; prediction
MeSH Terms: conditions — Sepsis; Hyperammonemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: Septic patients with positive microbial cultures.
- Group II: septic patients with negative microbial culture

SUMMARY:
Objectives: This study aims to determine the validity of hyperammonemia in predicting true sepsis compared to hyperlactemia in critically ill septic patients.

Background: Sepsis is associated with amino acid flux towards the liver, which increases the ammonia load. The combination of decreased clearance and increased load is thought to be the major cause of increased ammonia in sepsis.

Methodology: 60 septic patients were classified into 2 equal groups, Group I: Septic patients with positive microbial cultures. Group II: septic patients with negative cultures enrolled to obtain serum ammonia and lactic acid levels on admission and every six hours for three days. The primary outcome was to detect ammonia specificity and sensitivity in predicting sepsis in comparison to lactate. The secondary outcomes were need for mechanical ventilation, mortality, and length of stay (LHS) within the intensive care unit.

DETAILED DESCRIPTION:
Objectives: The study compares between non-cirrhotic hyperammonemia and hyperlactemia in predicting sepsis in critically ill septic patients.

The septic patients were classified into 2 equal groups, Group I: Septic patients with positive microbial cultures. Group II: septic patients with negative cultures enrolled to obtain serum ammonia and lactic acid levels on admission and every six hours for three days, to detect ammonia specificity and sensitivity in predicting sepsis in comparison to lactate. also, need for mechanical ventilation, mortality, and length of stay (LHS) within the intensive care unit were reported.

ELIGIBILITY:
Inclusion Criteria:

* adult patients aged 19-75 years old
* both sexes with severe sepsis and septic shock
* within the first 48 hours of ICU admission

Exclusion Criteria:

* Hepatic patients (cirrhotic, hepatitis),
* Renal failure, Ureterosigmoidostomy,
* Malignancy or on Chemotherapy,
* Pregnancy,
* Parenteral nutrition,
* Autoimmune diseases or Immunosuppressive illness, and
* Trauma

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with sepsis or septic shock
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Serum ammonia specificity and sensitivity in predicting sepsis in comparison to lactate | up to three days.
  Blood samples to obtain Serial ammonia and lactic acid levels

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia Faculty of Medicine, Shibin Elkoom, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No
it needs patient and institutional ethical committee approval